CLINICAL TRIAL: NCT04941027
Title: Evaluating Genetic Modifiers of Cutaneous Neurofibromas in Adults With Neurofibromatosis Type 1
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Johns Hopkins University (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Kavita Sarin, Assistant Professor of Medicine, Stanford University
Other Study IDs: 53000; MZ-0053000 (Other: OnCore); SPO: 200898 (Other Grant/Funding Number: Johns Hopkins University: PRIME NTAP)
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Neurofibromatosis 1
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Saliva samples will be collected from patients for genetic sequencing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main goal of this protocol is to develop a well-phenotyped genetic biobank to identify genetic variants associated with the heterogeneous clinical presentations of Neurofibromatosis Type 1 (NF1). This will allow for improve understanding of NF1 pathogenesis and more personalized disease management. The investigators will conduct a GWAS analysis to identify common genetic risk variants associated with the development of cutaneous neurofibromas.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 or older.
* NF type 1 diagnosed using clinical criteria.
* At least one neurofibroma present at time of enrollment.
* Patient able to read and understand consent form (or equivalent translation) and able to give consent.
* Patient able and willing to complete all study procedures.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants aged 40 or older that have been clinically diagnosed with NF1 and currently have neurofibromas present.
Sampling Method: Non-Probability Sample
Enrollment: 1046 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Determination of genetic variants associated with clinical presentations of NF1. | Day 1
  GWAS analysis will identify common genetic risk variants associated with the development of cutaneous neurofibromas in patients with NF1.

CONTACTS AND LOCATIONS:
Overall Officials: Kavita Sarin, MD PhD, Principal Investigator — Stanford University; Jaishri Blakely, MD, Principal Investigator — Johns Hopkins University; Carlos Romo, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University School of Medicine, Baltimore, California
  - Stanford University, Redwood City, California

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared indefinitely with collaborators after data is deidentified.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available as generated indefinitely.
Access Criteria: Data will be shared through secure REDCap database.